CLINICAL TRIAL: NCT04634604
Title: A Randomized Trial of Low-Dose Bevacizumab Versus Laser for Type 1 Retinopathy of Prematurity
Brief Title: A Randomized Trial of Low-Dose Bevacizumab vs Laser for Type 1 ROP
Acronym: ROP3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of feasibility to recruit.
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROP3; UG1EY011751 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab; Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Laser (Active Comparator): For infants randomized to laser treatment, it will be given in conjunction with a binocular indirect ophthalmoscope and an appropriate condensing lens, by a study-certified ophthalmologist experienced in the use of this equipment. The treating investigator will be certified as having sufficient experience with laser for ROP, and adequacy of laser treatment will be confirmed by expert review of photographs. Special laser precautions, as mandated by Occupational Safety and Health Administration (OSHA) and facility standards, will be followed.
  Interventions: Procedure: Laser
- Bevacizumab (Experimental): For infants randomized to bevacizumab, the Intravitreous bevacizumab 0.063 mg injection will be given no later than 2 days after the diagnosis of type 1 ROP. The ophthalmologist may choose to give the intravitreous injection in the operating room or at the bedside, with or without anesthesia, after consultation with the attending neonatologist. A binocular indirect ophthalmoscope with an appropriate condensing lens should be available, and the pupils should be dilated.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — For infants randomized to bevacizumab, the Intravitreous bevacizumab 0.063 mg injection will be given no later than 2 days after the diagnosis of type 1 ROP. The ophthalmologist may choose to give the intravitreous injection in the operating room or at the bedside, with or without anesthesia, after consultation with the attending neonatologist. A binocular indirect ophthalmoscope with an appropriate condensing lens should be available, and the pupils should be dilated.
  Other Names: Avastin
  Arms: Bevacizumab
Procedure: Laser — For infants randomized to laser treatment, it will be given in conjunction with a binocular indirect ophthalmoscope and an appropriate condensing lens, by a study-certified ophthalmologist experienced in the use of this equipment. The treating investigator will be certified as having sufficient experience with laser for ROP, and adequacy of laser treatment will be confirmed by expert review of photographs. Special laser precautions, as mandated by OSHA and facility standards, will be followed.
  Arms: Laser

SUMMARY:
This randomized clinical trial will compare retinal outcomes with low-dose intravitreous bevacizumab (0.063 mg) versus laser photocoagulation as treatment for infants with type 1 retinopathy of prematurity (ROP).

The study also will assess neurodevelopment, refractive error, visual acuity, and peripheral visual fields.

DETAILED DESCRIPTION:
Infants with type 1 ROP and no prior treatment for ROP will be randomly assigned (1:1) to treatment with either intravitreous bevacizumab 0.063 mg or peripheral retinal laser ablation. Study exams will be at weeks 1, 2, and 4 weeks, and at 2 and 4-months post-treatment (and re-treatment when indicated). Additional study exams will occur at adjusted age 6 months, 1 year, and then annually for 5 more years. Non-study examinations will be at clinician discretion and are likely to occur more often. The primary outcome will be treatment success, defined as no worsening of ROP 5-13 days after treatment (or re-treatment if indicated), no plus disease or severe neovascularization 2 weeks to 6 months after treatment (or re-treatment if indicated), and no unfavorable structural outcome (or prior scleral buckle or vitrectomy) at 6 months adjusted age. Important secondary outcomes include the number of re-treatments, extent of retinal vascularization, refractive error, neurodevelopment assessed by the Bayley-4 test, IQ and neuropsychiatric testing, visual acuity, visual fields, and systemic morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1251 grams
* Newly diagnosed (within 2 days) type 1 ROP in one or both eyes; meeting the following criteria:

  * Zone I, any stage ROP with plus disease, with retinal vessels or ROP in Zone II in any quadrant, or
  * Zone I, stage 3 ROP without plus disease, with retinal vessels or ROP in zone II in any quadrant or
  * Zone II, stage 2 or 3 ROP with plus disease

Exclusion Criteria:

* Previous treatment for ROP
* Stage 4 or 5 ROP in either eye
* All ROP in zone I in either eye (no retinal vessels or ROP extend into zone II in any quadrant)
* Either treatment could not be done within 2 days of diagnosis of type 1 ROP
* Investigator unwilling to randomize or parent unwilling to accept random assignment to either treatment
* Transfer to another hospital not covered by study-certified examiners anticipated within the next 4 weeks
* Active ocular infection or purulent nasolacrimal duct obstruction in either eye

One eye will be excluded, and other eye may be eligible, if either of the following are present:

* Visually significant ocular anomaly (e.g., cataract, coloboma)
* Opacity that precludes an adequate view of the retina

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Wallace, MD, MPH, Study Chair — Indiana University
Locations (35):
- United States (32):
  - Arizonia Pediatric Eye Specialists, Phoenix, Arizona
  - Arkansas Childrens Hospital/ University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Connecticut Childrens Medical Center, Farmington, Connecticut
  - The Emory Eye Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - U of Illinois at Chicago Eye and Ear Infirmary, Chicago, Illinois
  - University of Chicago, Hyde Park, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - UK Ophthalmology and Visual Sciences, The Eye Clinic, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Missouri- Columbia Mason Eye Institute, Columbia, Missouri
  - St. Louis University Ophthalmology, St Louis, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - New York Presbyterian David H Koch Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - Casey Eye Institute, Portland, Oregon
  - UPMC Children's Eye Center of Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Storm Eye Institute, Mt. Pleasant, South Carolina
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - University of Utah Moran Eye Center, Salt Lake City, Utah
  - Virginia Pediatric Eye Center, Norfolk, Virginia
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU - Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Yes In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- See also: PEDIG Public Website — http://www.pedig.net

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser | Bevacizumab
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Laser | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational Age
  weeks | 25 (1) | 24 (1) | 24 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Birth Weight [Mean (Standard Deviation); unit: grams] | 698 (122) | 670 (141) | 682 (129)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Rate At 6 Months Adjusted Age
Description: The primary objective for the randomized trial is to determine if infants with type 1 ROP treated with intravitreal bevacizumab (subsequently referred to as BV) have a treatment success rate determined at 6 months adjusted age that is non-inferior compared with infants treated with laser photocoagulation (subsequently referred to as LASER).
Time Frame: 6 Months Adjusted Age
Population: Study terminated due to lack of feasibility of recruitment. No analyses conducted due to lack of power for analysis given small sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Laser
Number analyzed (Participants) | 3 | 5
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study until study completion, up to 1 year (terminated early).
Arm/Group | Bevacizumab | Laser
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/9
Other Adverse Events (participants affected / at risk) | 4/7 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=7) | Laser (N=9)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Primary Apnea of premature newborns (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory insufficiency (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=7) | Laser (N=9)
Corneal edema (Eye disorders) | 1 (1) | 0 (0)
Esotropia (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 1 (2) | 0 (0)
Preretinal Hemorrhage (Eye disorders) | 0 (0) | 2 (3)
Retinal Hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bloody stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Electrolyte and fluid balance condition (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Viral Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Oxygen Saturations Low (Investigations) | 0 (0) | 1 (1)
Fractured Ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neurologic disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Primary apnea of premature newborns (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects which precluded statistical analysis. Active participants were released from study at time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT04634604/Prot_003.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04634604/SAP_001.pdf
  • Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT04634604/ICF_004.pdf